CLINICAL TRIAL: NCT06343870
Title: Pharmacokinetic, Clinical, Hormonal and Therapeutic Effects of the Use of Estradiol and Testosterone Hormonal Subdermal Implants in Women With Natural Menopause, Premature Ovarian Failure or Surgical Menopause Due to Cervical Cancer.
Brief Title: Estradiol and Testosterone Subdermal Implants for Menopause Treatment (ESTIME)
Acronym: ESTIME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Edmund Baracat, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESTIME
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Menopause; Testosterone Deficiency; Estrogen Deficiency
Keywords: menopause; estrogen; testosterone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Active Comparator): Subdermal implant-bioabsorbable testosterone pellet (100 mg of testosterone)
  Interventions: Drug: testosterone pellet (100 mg)
- Placebo (Placebo Comparator): Subdermal implant-bioabsorbable placebo pellet (cholesterol)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: testosterone pellet (100 mg) — Intervention arm: Subdermal implant-bioabsorbable testosterone pellet (100 mg of testosterone)
  Other Names: testosterone subdermal implant
  Arms: Testosterone
Drug: Placebo — Pellet of cholesterol (placebo)
  Arms: Placebo

SUMMARY:
Estrogen and androgen deficiencies negatively impact the quality of life of women at different stages of life, especially after menopause. New modalities and new therapeutic alternatives have been researched. Parenteral administration of estradiol and testosterone could be effective to treat symptoms secondary to estrogen and androgen deficiencies and minimize these adverse events. This study evaluates the efficiency of subdermal implant-bioabsorbable use in women with menopausal symptoms associated with secondary estrogen and androgen deficiencies in women with natural menopause, premature ovarian failure or surgical menopause due to cervical cancer. Pharmacokinetic, biochemical, metabolic, thromboembolic and hormonal data will be evaluated, as well as the effects on quality of life, menopausal symptoms and sexual function after treatment.

DETAILED DESCRIPTION:
The clinical study will be carried out on 140 women, who will be divided into three groups: (1) postmenopausal women with menopausal and sexual symptoms (n=60); (2) women with premature ovarian failure (n=40); (3) women with cervical cancer undergoing abdominal hysterectomy with bilateral adnexectomy, with menopausal and sexual symptoms (n=40).

All participants will answer questionnaires to assess quality of life, menopausal symptoms and sexual function. All participants will undergo general physical and gynecological examinations, as well as hormonal, biochemical, thromboembolic and imaging tests.

The study will last six months. The included participants will undergo the following visits: inclusion (post-selection) and 1, 3 and 6 months after implant insertion. For the pharmacokinetic study, blood samples will be collected at the following periods: inclusion (before implant placement) and after 1h, 2h, 3h, 6h and 12h; one week, two weeks and one month after placement, and then monthly until six months after implant insertion, to evaluate serum levels of Luteinizing hormone, Follicle stimulating hormone, estradiol, estrone, total testosterone and sex hormone-binding globulin.

Clinical, biochemical, hormonal and therapeutic parameters will be evaluated before placement (inclusion) and after 3 and 6 months. The Mann Whitney test will be applied to evaluate differences between measurements and the chi-square test will be applied to analyze the proportions of improvement between groups before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* menopause time of 2 to 6 years;
* Body Mass Index between 25 and 30 kg/m2;
* women hysterectomized and ovariectomized due to cervical cancer;
* women with premature ovarian failure and under 40 years of age;
* active sex life;
* absence of severe depression and anxiety, confirmed by evaluation using the Beck (specific for depression) and Beck (specific for anxiety) questionnaires.

Exclusion Criteria:

* disabling illnesses;
* use of medications that inhibit sexual desire;
* inability to answer the questionnaires;
* altered routine exams and comorbidities:

  * Severe hypertension with Blood Pressure measurement > 160 x 90 mmHg in two measurements
  * clinical or subclinical thyroid dysfunction with Thyroid-stimulating hormone > 4 mIU/L
  * dyslipidemia - fasting triglyceride level > 400 mg/dL
  * presence of occult blood in feces
  * hyperprolactinemia (>29ng/mL)
  * fasting blood glucose > 100 mg/dL
  * presence of osteopenia or osteoporosis
  * BIRADS classification greater than or equal to 3 on mammography
  * presence of endometrial echo > 4mm on transvaginal ultrasound
  * presence of changes in oncotic colpocytology
* diagnosis after psychological screening of moderate to severe anxiety/depression.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate hormonal, metabolic thromboembolic and clinical effects on climacteric symptoms | 6 months
  evaluate concentration in serum of luteinizing hormone, follicle stimulating hormone, estradiol, estrone, total testosterone and sex hormone-binding globulin.

SECONDARY OUTCOMES:
Evaluate response in quality of life and sexual function | 6 months
  Evaluate response on vulvovaginal atrophy and genitourinary syndrome of menopause, hormonal and metabolic effects on climacteric symptoms, using the Kupperman Menopausal Index; response in quality of life and sexual function; hormonal and metabolic effects;

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Baracat, PhD, Principal Investigator — Instituto do Coracao
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lev-Sagie A. Vulvar and Vaginal Atrophy: Physiology, Clinical Presentation, and Treatment Considerations. Clin Obstet Gynecol. 2015 Sep;58(3):476-91. doi: 10.1097/GRF.0000000000000126. PMID 26125962
- [Background] Nelson HD. Menopause. Lancet. 2008 Mar 1;371(9614):760-70. doi: 10.1016/S0140-6736(08)60346-3. PMID 18313505
- [Background] Calleja-Agius J, Brincat MP. The urogenital system and the menopause. Climacteric. 2015;18 Suppl 1:18-22. doi: 10.3109/13697137.2015.1078206. PMID 26366796
- [Background] The NAMS 2020 GSM Position Statement Editorial Panel. The 2020 genitourinary syndrome of menopause position statement of The North American Menopause Society. Menopause. 2020 Sep;27(9):976-992. doi: 10.1097/GME.0000000000001609. PMID 32852449
- [Background] Suhonen SP, Allonen HO, Lahteenmaki P. Sustained-release estradiol implants and a levonorgestrel-releasing intrauterine device in hormone replacement therapy. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):562-7. doi: 10.1016/0002-9378(95)90573-1. PMID 7856686
- [Background] Kingsberg S, Althof SE. Evaluation and treatment of female sexual disorders. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20 Suppl 1:S33-43. doi: 10.1007/s00192-009-0833-x. PMID 19440781
- [Background] Brincat M, Magos A, Studd JW, Cardozo LD, O'Dowd T, Wardle PJ, Cooper D. Subcutaneous hormone implants for the control of climacteric symptoms. A prospective study. Lancet. 1984 Jan 7;1(8367):16-8. doi: 10.1016/s0140-6736(84)90183-1. PMID 6140343